CLINICAL TRIAL: NCT00515801
Title: Effect of a Sulfonylurea Compound on the Glucagon Response to Insulin-induced Hypoglycemia in Type 1 Diabetes Mellitus
Brief Title: Sulfonylurea Effects on Glucagon Regulation During Hypoglycemia in Type 1 DM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EKBB 57/07 SB
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes mellitus type 1; hypoglycemia; sulfonylurea; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glyburide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Glibenclamide 5 mg tablets
  Interventions: Drug: glibenclamide
- B (Placebo Comparator): placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glibenclamide — glibenclamide 15 mg single dose
  Other Names: Daonil 5 mg pills
  Arms: A
Drug: placebo — placebo capsules, single dose
  Arms: B

SUMMARY:
We aim to demonstrate that oral administration of glibenclamide stimulates pancreatic glucagon secretion during hypoglycemia in insulin-deficient (C-peptide negative) patients with type 1 diabetes when compared to type 1 diabetic patients with residual insulin secretion (C-peptide positive).

DETAILED DESCRIPTION:
The glucagon response during insulin induced hypoglycemia and rate of glucose recovery will be monitored in 10 C-peptide positive and 10 C-Peptide negative patients with type 1 DM following the application of glibenclamide and placebo in a randomized, single-blind, cross-over study.

Cognitive function during hypoglycemia with and without glibenclamide pretreatment will be a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 50 years
* Patients diagnosed with C-peptide negative diabetes type 1 (C-peptide <200 pmol/L 6 min after 1 mg glucagon i.v. at plasma glucose concentrations between 5 and 11 mmol/l)
* Patients diagnosed with C-peptide positive diabetes type 1 (C-peptide > 500 pmol/l 6 min after 1 mg glucagon i.v. at plasma glucose concentrations between 5 and 11 mmol/l)
* Stable metabolic control; HbA1c levels <8.0 % and without episodes of antecedent severe hypoglycemias in the past four weeks

Exclusion Criteria:

* Patients treated with medications potentially interfering with glucose metabolism, such as systemic steroids, immunosuppressive drugs (cyclosporine, tacrolimus, sirolimus), highly active antiretroviral therapy
* History coronary artery disease
* History of epilepsy or seizures
* Current smokers
* Any significant or unstable hepatic, cardiac, pulmonary, renal, neurological, musculoskeletal, hematological or endocrine disease.
* Pregnant or breast feeding women
* Woman of childbearing potential not using a reliable method of birth control such as oral contraceptives or IUD.
* Subjects refusing or unable to give written informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-06

PRIMARY OUTCOMES:
plasma glucagon concentrations during insulin induced hypoglycemia with and without glibenclamide pretreatment | cross-sectional

SECONDARY OUTCOMES:
rate of glucose recovery following insulin induced hypoglycemia with and without glibenclamide pretreatment | cross-sectional
cognitive function during insulin induced hypoglycemia with and without glibenclamide pretreatment | cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bilz, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Seelig E, Bilz S, Keller U, Meienberg F, Christ-Crain M. Concentrations of the stress hormone copeptin increase upon hypoglycaemia in patients with type 1 diabetes dependent of hypoglycaemia awareness. PLoS One. 2013 Aug 30;8(8):e72876. doi: 10.1371/journal.pone.0072876. eCollection 2013. PMID 24023652